CLINICAL TRIAL: NCT06462924
Title: Feasibility of Gadolinium Contrast Reduced Brain MRI: the Potential of Deep Learning
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: DeepMeds (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DG53024
Record Dates: First submitted 2024-05-30; First posted 2024-06-17 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Artificial Intelligence; Deep Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DeepGad (Experimental): The dataset comprises a total of 500 patients, with 300 patients used for model training and 200 patients reserved for model testing. Each patient had approximately 350 2D brain slices of the coregistered 3D volumes excluding the five slices at the base and five slices at the top of the acquired volume due to their low signal-to-noise ratio (SNR). For robustness and to avoid overfitting, standard DL data augmentation techniques consisting of eight types of transformations were applied to each case in the training set.
  Interventions: Device: DeepGad

INTERVENTIONS:
Device: DeepGad — Using the pre-contrast and low-dose Contrast-Enhanced Magnetic Resonance (CE-MRI) images as input and the true full-dose CE-MRI images as the ground truth. the Cycle GAN deep network (DeepGad), was trained to reconstruct the full-dose CE-MRI images from low-dose CE-MRI images.

SUMMARY:
MRI scans were performed using 3 different 1.5T scanners with an eight-channel head coils. Following a 3D pre-contrast T1w scan, a low-dose contrast-enhanced 3D T1w scan was obtained using 20% (0.02 mmol/kg) of the standard dosage of gadoterate meglumine.

The subjects were immediately administered the remaining 80% (0.08 mmol/kg) of the contrast agent to reach the standard dose of 0.1 mmol/kg, which served as a training ground truth for further quantitative assessment. All three acquisitions were performed during a single imaging session, with no additional gadolinium dose administered above the standard protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indications for imaging with a contrast-enhanced 3D-T1w MRI sequence including tumor suspicion, postoperative tumor follow-up, multiple sclerosis, routine brain imaging, etc.,
2. no plan for dynamic contrast administration or deviation from the standard dose of 0.1 mmol/kg body weight (e.g., sella imaging, magnetic resonance angiography),
3. no clinical contraindications to imaging prolongation (i.e., emergency, poor patient condition).

Exclusion Criteria:

1. prominent image artifacts,
2. incomplete study sequences (e.g., early termination)
3. errors related to contrast agent administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Image quality | 1 Day After MRI session
  Image quality using a 5-point Likert scale covering 1 (none), 2 (poor), 3 (moderate), 4 (good), and 5(excellent) ratings
Vessel conspicuity | 1 Day After MRI session
  (0) no normal vessels observed, (1) significant decrease in conspicuity with potential impact on diagnosis, (2) mild decrease in conspicuity with unlikely impact on diagnosis, (3) normal conspicuity, (4) mild increase in conspicuity with unlikely impact on diagnosis, and (5) significant increase in conspicuity with potential impact on diagnosis.

SECONDARY OUTCOMES:
Enhancement pattern | 1 Day After MRI session
  (a) no enhancement, (b) homogeneous enhancement, (c) heterogeneous enhancement, (d) ring enhancement, (e) linear enhancement, and (f) other enhancement.

IPD SHARING:
Plan to Share IPD: No